CLINICAL TRIAL: NCT06331052
Title: 3-D Tractography Focused Ultrasound Ablation for Essential Tremor
Brief Title: 3-D Tractography FUS Ablation for Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Texas Tech University Health Sciences Center, El Paso (Other); University of Pittsburgh (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-2431; 1R01NS125386-01 (NIH)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 3-D Tractography Vim FUSA (Experimental): Twenty-four consecutive essential tremor (ET) participants undergoing Vim FUSA using 3-D tractography will be assessed at baseline and Month 3.
  Interventions: Device: MR-guided Focused Ultrasound Ablation

INTERVENTIONS:
Device: MR-guided Focused Ultrasound Ablation — 3-D tractography Vim-FUSA -D tractography Vim-FUSA will be carried out as follows: (a) head shaving and placement of the stereotactic frame (Integra radionics frame, Integra Lifesciences, NJ, USA) secured to the skull with transcutaneous screws; (b) positioning on the procedure table and placement of the ultrasound transducer; (c) acquisition of conventional magnetic resonance (MR) imaging and co-registration with the CT head and 3-D tractography imaging acquired pre-surgically; (d) exploration of the target area with subtherapeutic sonications; (e) intraoperative monitoring with clinical testing of tremor and side effects with a standardized protocol. (f) Therapeutic sonications in the target area to deliver definitive ablation followed by clinical testing of tremor and side effects with a standardized protocol as described in section (e).
  Other Names: 3-D Tractography

SUMMARY:
The investigators propose to advance Vim-FUSA (Ventral Intermediate Nucleus - Focused Ultrasound Ablation) with the support of 3-D tractography, a neuroimaging technique to visually represent nerve tracts within the brain. The investigators hypothesize that 3-D tractography Vim-FUSA will improve the Vim ablation compared to standard Vim-FUSA and prove safe and feasible in the clinical setting. The investigators also hypothesize that intraoperative magnetic resonance (i-MR) monitoring will differentiate ablated tissue from immediate perilesional edema and accurately predict the Vim-FUSA clinical outcomes.

DETAILED DESCRIPTION:
Essential tremor (ET) is a common neurological disorder and a leading cause of functional and psychological disabilities that can be difficult to suppress with oral medications, many of which have considerable side effects limiting adequate dosing. As a result, up to 20% of ET patients cannot achieve satisfactory control of their symptoms and must consider interventional options. Focused ultrasound ablation (FUSA) of the ventral intermediate nucleus (Vim) is an FDA-approved and Medicare-reimbursed procedure for ET resistant to medications that can selectively ablate the brain area associated with tremor without the need for surgical incisions or anesthesia. The success of Vim-FUSA depends on the ability to accurately ablate 70% of the Vim volume without lesioning neighboring structures, a goal that is complicated by technical challenges in three critical phases of the procedure: planning (identifying the Vim location and extension); delivery (ablating the Vim volume with adequate accuracy); and monitoring (confirming Vim ablation with reliable intraoperative imaging). The investigators propose to advance Vim-FUSA with the support of 3-D tractography, a neuroimaging technique to visually represent nerve tracts within the brain. The investigators hypothesize that 3-D tractography Vim-FUSA will improve the Vim ablation compared to standard Vim-FUSA and prove safe and feasible in the clinical setting. The investigators also hypothesize that intraoperative magnetic resonance (i-MR) monitoring will differentiate ablated tissue from immediate perilesional edema and accurately predict the Vim-FUSA clinical outcomes. Aim 1. Estimate and characterize the improvement in Vim ablation achieved with 3-D tractography Vim-FUSA vs. standard Vim-FUSA in an experimental controlled animal study. Through an experimental animal study, the investigators will characterize the Vim ablation delivered with 3-D tractography Vim-FUSA in one hemisphere (experimental group) vs. standard Vim-FUSA in the opposite hemisphere (control group). Aim 2. Test safety, feasibility, and preliminary efficacy, and estimate effect size of 3-D tractography Vim-FUSA in a phase-II, two-groups, pre-post interventional human study. In a human study, the investigators will test the safety and feasibility of ablating 70% of the Vim volume while checking for side effects with intraoperative clinical testing. Tremor assessments will be videotaped at baseline and 12 weeks and compared, in a blinded fashion, with age-sex matched controls randomly selected from the video repository of the two FDA-regulated studies of standard Vim-FUSA at baseline and 12 weeks. Aim 3 (Exploratory). Assess the accuracy of i-MR in differentiating tissue ablation from immediate perilesional edema and its utility in predicting Vim-FUSA clinical outcomes. In the experimental animal study, the investigators will estimate and compare the accuracy of conventional and non-conventional i-MR in differentiating tissue necrosis from perilesional edema. In the interventional human study, the investigators will evaluate the utility of i-MR in predicting Vim-FUSA clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe ET agreed upon by at least two movement disorder trained physicians
* Symptoms refractory to at least two medications
* Stable medication regimen for at least 4 weeks prior to screening
* Willing and able to participate in all follow-up visits
* Willing and able to undergo MR imaging.

Exclusion Criteria:

* Uncontrolled hypertension
* Medically unstable coronary artery disease
* Coagulopathy, anticoagulant therapy, or inability to temporarily stop any antithrombotic medication
* Tremor disorders other than ET
* Unwilling or unable to undergo tremor surgery while awake
* Significant and non-correctible motion artifact in imaging
* Pregnant at the time of enrollment or preoperative evaluation
* Dementia
* History of psychosis
* History of drug or alcohol abuse
* Prior brain surgery such as Vim-FUSA, deep brain stimulation, and gamma knife thalamotomy
* Botulinum toxin injection in the tremor-impacted areas three months prior to the baseline assessment and until 3-months after Vim-FUSA
* Skull density ratio lower than 0.4
* Does not qualify for FDA-approved clinical use based on current FDA labeling
* Any significant issue raised by the neurologist or neurosurgeon that may compromise participant safety or potentially interfere with study interpretation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants without Side Effects | during the surgical procedure
  Feasibility is defined as the ability to complete the procedure without side effects.
Absolute Change in Tremor | Baseline, Month 3
  The absolute change from baseline to Month 3 follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and 3 Months used to calculate absolute change from baseline and averaged across subjects. High absolute change from baseline is better (shows improvement).
Relative Change in Tremor | Baseline, Month 3
  The relative change from baseline to Month 3 follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and 3 Months used to calculate relative change from baseline and averaged across subjects. High relative change from baseline is better (shows improvement).

SECONDARY OUTCOMES:
Number of Participants with Procedure-Related Side Effects | 3 months after the surgical procedure
  Prevalence and severity of procedure-related side effects measured by the following: ataxia (SARA), speech disturbance (VHI), sensory loss (SWME), muscle weakness (MRC)
Relative Change in Tremor-Related Quality of Life | 3 months after the surgical procedure
  The Quality of Life Essential Tremor Questionnaire (QUEST) will be used to assess tremor-related quality of life. QUEST has scores ranging from 0 to 100 with higher scores indicating worse disability.
Number of Participants Who Are Satisfied with Treatment | 3 months after the surgical procedure
  Measured using a single question asking about patient satisfaction ranging from 1 to 5 with higher scores indicating higher satisfaction.

OTHER OUTCOMES:
Change in Tremor Based on Video Assessment | Baseline, during the surgical procedure
  Upper extremity tremors will be measured by video recording using i-Phone set-up.
Change in Gait Based on Video Assessment | Baseline, during the surgical procedure
  Gait will be measured by video recording using i-Phone set-up.

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor Krishna, MD, Principal Investigator — University of North Carolina at Chapel Hll
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC REB and an executed data use/sharing agreement with UNC.